CLINICAL TRIAL: NCT03769480
Title: Investigation of the Relationship Between Pulmonary Function and Muscle Strength in Athletes With Disability
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Bihter Aslanyurek, Principal Investigator, Ankara Yildirim Beyazıt University
Other Study IDs: 2
Record Dates: First submitted 2018-11-29; First posted 2018-12-07 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Disabilities Multiple
Keywords: Athletes; Disability; Respiratory Function; Core Muscles; Sport
MeSH Terms: conditions — Respiratory Aspiration | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Study Group=Athletes with Disability
  Interventions: Other: Muscle strength evaluation and Respiratory function Tests
- Control Group: Control Group=Healthy Athletes
  Interventions: Other: Muscle strength evaluation and Respiratory function Tests

INTERVENTIONS:
Other: Muscle strength evaluation and Respiratory function Tests — Muscle strength evaluation and Respiratory function Tests

SUMMARY:
To investigate the relationship between respiratory function and core muscles strength in athletes with disabilities and compare with healthy athletes.

DETAILED DESCRIPTION:
The determination of parameters affecting the performance of high performance athletes that are effective in performance is very important to determine the physical performance potential. The body is a kinetic chain and core muscles play an important role in this chain. The relationship between the performance ability of the athletes and the relationship between the core muscles and performance abilities and respiratory function is extremely important. Different functional classifications caused by different barriers (physical, mental or visual) in many paralympic branches affect physical training because it is directly related to the classification, performance and training adaptations of an athlete. Determining the parameters that affect the respiratory function of paralympics is very important to develop a training program with strategies that can affect the physical performance of athletes and thus to achieve the desired results in training and competitions. Therefore, the aim of this study was to investigate the relationship between respiratory muscle strength and core muscle strength in paralympic athletes (athletes with disability).

ELIGIBILITY:
Inclusion Criteria:

* Being professional athletes for at least three years.

Exclusion Criteria:

* Having any lumbar injuries in the last three months,
* Having systemic problems other than their disabilities(for athletes with disabilities),
* Having any disability related to vision and hearing,
* Acute or chronic respiratory infection,
* Spinal cord injury level up to the innervation of the abdominal muscles (for paraplegic athletes).

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study group is Athletes with disabilities.
  The control group is the same sport branches but healthy athletes without any disabilites
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
FVC (the rate of normal value by the spirometer device) | 2 days
  Functional vital capacity: will evaluate by the rate of normal value by the spirometer device (Pony FX Cosmed device)
FEV1 ( the rate of normal value by the spirometer device) | 2 days
  First second Forced Expiratory Volume:will evaluate by the rate of normal value by the spirometer device (Pony FX Cosmed device)
Muscle strength (Abdominal Flexor Muscle Strength: will evaluate as Newtonmeter (Nm) by isokinetic device) | 2 days
  Abdominal Flexor Muscle Strength: will evaluate as Newtonmeter (Nm) by isokinetic device (IsoMed 2000, trunk attachment).
Muscle strength (Abdominal Exstansor Muscle Strength: will evaluate as Newtonmeter (Nm) by isokinetic device) | 2 days
  Abdominal Extensor Muscle Strength: will evaluate as Newtonmeter (Nm) by isokinetic device (IsoMed 2000, trunk attachment).
Muscle strength (Abdominal right rotator Muscle Strength: will evaluate as Newtonmeter (Nm) by isokinetic device) | 2 days
  Abdominal right rotator Muscle Strength: will evaluate as Newtonmeter (Nm) by isokinetic device (IsoMed 2000, trunk attachment).
Muscle strength (Abdominal left rotator Muscle Strength: will evaluate as Newtonmeter (Nm) by isokinetic device) | 2 days
  Abdominal left rotator Muscle Strength: will evaluate as Newtonmeter (Nm) by isokinetic device (IsoMed 2000, trunk attachment).

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Kocahan, Dr, Study Chair — The Ministry of Youth and Sports, Sports General Directorship, Ankara, Turkey
Locations (1):
- Bihter Akınoğlu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The participants all is national team. Because we can not share the data